CLINICAL TRIAL: NCT05885763
Title: A Phase 1, Single-arm, Open-label Study to Evaluate the Pharmacokinetics and Safety of Intravenous Difelikefalin in Adult Chinese Subjects on Haemodialysis
Brief Title: Pharmacokinetics of Intravenous Difelikefalin in Chinese Adult Subjects on Haemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-CHINA-101; JXHL2101166 (Other: Center for Drug Evaluation (CDE) China)
Record Dates: First submitted 2023-05-17; First posted 2023-06-02 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease on Hemodialysis
Keywords: Difelikefalin; Pharmacokinetics
MeSH Terms: interventions — difelikefalin

STUDY DESIGN:
Intervention Model Description: A Single-arm, Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1-week, single arm, open label treatment phase (Experimental)
  Interventions: Drug: Difelikefalin Injection

INTERVENTIONS:
Drug: Difelikefalin Injection — Participants receive Difelikefalin three times a week (0,5 micrograms/kg dry body weight). Difelikefalin is administered by intravenous bolus injection into the venous line of the dialysis circuit at the end of each dialysis.

SUMMARY:
This is a Phase 1, single-arm, open-label study to evaluate the safety, PK, and tolerability of a repeated (3 times weekly) dose of difelikefalin administered as IV bolus injections to adult Chinese HD subjects. Treatment period is one week and there is a safety follow-up period of 1 week.

DETAILED DESCRIPTION:
This is a Phase 1, single-arm, open-label study to evaluate the safety, PK, and tolerability of a repeated (3 times weekly) dose of difelikefalin administered as IV bolus injections to adult Chinese HD subjects.

Total study duration for a single subject is up to 5 weeks including a screening period of up to 3 weeks, a treatment period of 1 week, and a safety follow-up period of 1 week.

The duration of PK sampling is 12 days.

The primary objective of the study is to evaluate the PK profile of a repeated (3 times weekly) dose of difelikefalin in Chinese HD subjects over a 1-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease (ESRD) subjects who have been on HD for at least 3 months before enrolment in the study and are currently on HD 3 times per week.
* Subjects with a prescription dry body weight between 40 and 100 kg, inclusive.
* If female, is not pregnant, or nursing
* If female:

  1. Is surgically sterile; or
  2. Has been amenorrhoeic for at least 1 year and is over the age of 55 years; or
  3. Has a negative serum pregnancy test within 7 days before first dose of investigational product, and agrees to use adequate contraceptive precautions (e.g., hormonal contraceptives, barrier with spermicide, intrauterine device, vasectomised partner, or abstinence) from the time of informed consent until 7 days after the last dose of investigational product.
* If male, agrees not to donate sperm from the first dose of investigational product administration (Day 1) until 7 days after last dosing, and agrees to use a condom with spermicide or abstain from heterosexual intercourse during the study until 7 days after the last dose of investigational product.

Exclusion Criteria:

* Planned or anticipated to receive a kidney transplant during the study.
* Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) greater than 2.5 × the reference upper limit of normal (ULN), or bilirubin (total) greater than 4 × the ULN at screening.
* Subjects with severe hepatic impairment (Child-Pugh Class C).
* Known history of allergic reaction to opiates such as hives. Note: Side effects related to the use of opioids such as constipation or nausea would not exclude the subjects from the study.
* Subject has known hypersensitivity to the study intervention or any component of the investigational product formulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milica Enoiu, PhD, Study Director — Vifor Pharma Group
Locations (4):
- China (4):
  - Investigator Site 1, Beijing
  - Investigator Site 2, Beijing
  - Investigator Site 3, Beijing
  - Investigator Site 4, Shijiazhuang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 30
Region of Enrollment [Number; unit: participants]
  China | 30

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - Cmax - Dose 1
Description: Cmax = Maximum (peak) observed plasma concentration
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
ng/mL | 3.70 (33.1)

2. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - Tmax - Dose 1
Description: Tmax = Time to reach maximum observed plasma concentration
Time Frame: 1 week
Measure: Median (Full Range); unit: Hours
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
Hours | 0.08 [0.05 to 0.98]

3. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - AUC0-t - Dose 1
Description: AUC0-t = Area under the concentration-versus-time curve (AUC) from time zero to time "t"
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
h*ng/mL | 48.3 (27.6)

4. Primary Outcome: AUCinf - Dose 1
Description: AUCinf = AUC from time zero to infinity
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
h*ng/mL | 63.2 (43.9)

5. Primary Outcome: AUCextrap(%) - Dose 1
Description: AUCextrap(%) = percentage of AUCinf based on extrapolation
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
percentage | 23.5 (49.3)

6. Primary Outcome: t½ - Dose 1
Description: t½ = elimination half-life
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
Hours | 22.2 (36.4)

7. Primary Outcome: Clearance - Dose 1
Description: Clearance = the volume of blood or plasma that can be freed of a specified constituent in a specified time by its excretion into the urine through the kidneys
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/H
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
L/H | 0.510 (43.6)

8. Primary Outcome: Vz - Dose 1
Description: Vz = volume of distribution
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 30
L | 16.3 (20.4)

9. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - Cmax - Dose 3
Description: Cmax = Maximum (peak) observed plasma concentration
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
ng/mL | 4.23 (23.8)

10. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - Tmax - Dose 3
Description: Tmax = Time to reach maximum observed plasma concentration
Time Frame: 1 week
Measure: Median (Full Range); unit: Hours
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
Hours | 0.08 [0.05 to 0.57]

11. Primary Outcome: Evaluation of the PK Profile of Difelikefalin - AUC0-t - Dose 3
Description: AUC0-t = Area under the concentration-versus-time curve (AUC) from time zero to time "t"
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
h*ng/mL | 65.6 (33.8)

12. Primary Outcome: AUCinf - Dose 3
Description: AUCinf = AUC from time zero to infinity
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
h*ng/mL | 77.6 (48.0)

13. Primary Outcome: AUCextrap(%) - Dose 3
Description: AUCextrap(%) = percentage of AUCinf based on extrapolation
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
percentage | 15.1 (61.4)

14. Primary Outcome: t½ - Dose 3
Description: t½ = elimination half-life
Time Frame: 1 week
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
Number analyzed (Participants) | 29
Hours | 25.0 (37.7)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported until the last study visit (up to 5 weeks) and Serious AEs (SAEs) until 30 days after the last study visit (up to 10 weeks).
Description: The SAE reporting period begins at the time the ICF is signed by the subject. The SAE reporting period ends 30 days following the last study visit. After last study visit, SAEs that comes to the attention of the Investigator must be reported to the CRO/Sponsor and will be documented in the safety database of the Sponsor only and not in eCRF. A rationale for the assessment of a causal relationship must be provided by the Investigator.
Arm/Group | 1-week, Single Arm, Open Label Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-week, Single Arm, Open Label Treatment Phase (N=30)
Abscess limb (Skin and subcutaneous tissue disorders) | 1 (1) — One subject discontinued the study, due to a pre-treatment SAE of abscess limb after receiving only 1 dose of study drug
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-week, Single Arm, Open Label Treatment Phase (N=30)
Paraesthesia (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT05885763/Prot_SAP_000.pdf